CLINICAL TRIAL: NCT02562287
Title: A Randomized Controlled Trial to Evaluate the Effectiveness of Clozapine Versus Olanzapine, Quetiapine or Risperidone in Treatment Resistant Bipolar Disorder
Brief Title: Clozapine Versus Other Atypical Antipsychotics for Bipolar Disorder
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Pedro Vieira da Silva Magalhães, Professor of Psychiatry, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 32356214200005327
Record Dates: First submitted 2015-08-11; First posted 2015-09-29 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Clozapine; Risperidone; Olanzapine; Quetiapine Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clozapine (Experimental): Clozapine, P.O., flexible dose, for up to 6 months
  Interventions: Drug: Clozapine
- Risperidone, olanzapine or quetiapine (Active Comparator): Risperidone, olanzapine or quetiapine, according to clinical indication, flexible dose, for up to 6 months
  Interventions: Drug: Risperidone; Drug: Olanzapine; Drug: Quetiapine

INTERVENTIONS:
Drug: Clozapine — Flexible dosage, with up-titration according to standard schedules employed for schezophrenia
  Other Names: Clozaril
  Arms: Clozapine
Drug: Risperidone — Risperidone, in a flexible dosage
  Other Names: Risperdal
  Arms: Risperidone, olanzapine or quetiapine
Drug: Olanzapine — Olanzapine, flexible dosage
  Other Names: Zyprexa
  Arms: Risperidone, olanzapine or quetiapine
Drug: Quetiapine — Quetiapine, flexible dosage
  Other Names: Seroquel
  Arms: Risperidone, olanzapine or quetiapine

SUMMARY:
The clinical use of clozapine has been an unequivocal advance in the treatment of schizophrenia, a chronic and severe mental illness. A wealth of clinical data demonstrates it offers enhanced efficacy on both positive and negative symptomatology, improving cognition, functioning and quality of life. It is also associated with improved compliance and a continued efficacy in long-term treatment that can be translated into a reduction of suicidality and all-cause mortality. Because of preclinical evidence that it modulates neuroplasticity and prefrontal cortex connectivity, clozapine may be an interesting strategy for further severe psychotic illnesses. Nevertheless, even considering the growing use of other atypical antipsychotics in the management of bipolar disorder, a role for clozapine has been poorly defined. The clinical evidence-base for its use in this condition is largely based on uncontrolled naturalistic trials and retrospective studies and chart reviews. Several of these have supported clozapine's efficacy in treatment-resistant bipolar disorder. Possibly because of clozapine's profile of adverse effects and lack of interest from pharmaceutical companies, only two randomized trials have examined its effectiveness. Both suggest clinically relevant antimanic and mood-stabilizing properties. Therefore, the primary objective of this trial is to determine the effectiveness of clozapine for treatment-resistant bipolar disorder. Secondary objectives include examining the effects of treatment with clozapine on cognition and functioning of patients with bipolar disorder. Tolerability and safety of long-term clozapine use will also be examined. To that end, the investigators will conduct a clinical trial with 54 patients with a history of treatment resistance. Patients will be randomized to either open-label treatment with clozapine, in combination with lithium or valproate, or open-label treatment with an atypical antipsychotic with consistent evidence of efficacy in the treatment of bipolar disorder (olanzapine, quetiapine or risperidone), also in combination with lithium or valproate. Patients will be followed for one-year and time to all-cause treatment failure will be the primary outcome measure. It is the belief of the investigators that this study will generate meaningful clinical data of tremendous importance to validate clozapine as a legitimate treatment option for treatment-resistant bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV Bipolar I Disorder;
* having had a mood episode within the preceding year; DSM-IV rapid cyclers will be permitted to participate in this study;
* males or females between 18 and 65 years of age;
* ongoing illness symptoms including significant functional impairment;
* documented history of treatment resistance, defined as persistent symptoms despite simultaneous, adequate treatment with at least two medications: one mood stabilizer (lithium or valproate) + antipsychotic OR two mood stabilizers (at least one of them being lithium or valproate).
* each patient must have a level of understanding sufficient to agree to all the tests required by the protocol and must sign an informed consent document

Exclusion Criteria:

* patients with onset of illness after age 40 or illness resulting from secondary causes
* women who are pregnant or breastfeeding, or not using adequate contraception
* unstable medical illnesses
* clinically significant abnormal laboratory tests
* current active alcohol or substance abuse
* severe personality disorders
* contraindication to the use of clozapine or previous treatment with clozapine

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2015-10; Primary Completion 2019-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Functioning according to Functioning Assessment Short-Test | 6 month follow up
  Global functioning according to Functioning Assessment Short-Test

SECONDARY OUTCOMES:
Time to all-cause treatment failure | Six months
  Include drug treatment (commencement of a new drug, restarting of a discontinued drug, or increasing the investigational drug dose in response to an emergent mood episode), admission to hospital or withdrawal from study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: PEDRO V MAGALHAES, M.D., Ph.D., Principal Investigator — Hospital de Clínicas de Porto Alegre / Universidade Federal do Rio Grande do Sul
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil